CLINICAL TRIAL: NCT00047255
Title: A Multicenter Phase III Randomized Trial Comparing Docetaxel (Taxotere) and Trastuzumab (Herceptin) With Docetaxel (Taxotere), Carboplatin and Trastuzumab (Herceptin) as First Line Chemotherapy for Patients With Advanced Breast Cancer Containing the HER2 Gene Amplification
Brief Title: Docetaxel and Trastuzumab With or Without Carboplatin in Treating Women With HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257580; UCLA-0109024 (Other: UCLA IRB); BCIRG-007 (Other: UCLA)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herceptin plus docetaxel (Experimental): Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose administered by IV infusion over 90 minutes, Day 2: Docetaxel (T) 100 mg/m2 by IV infusion over 30 minutes, Day 8: (H) 2mg/kg administered by IV infusion over 30 minutes, Day 15: 2mg/kg administered by IV infusion over 30 minutes.
  Subsequent cycles: Day 1: (T) 100mg/m2 as 1 hour IV infusion given every 3 weeks, followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes.
  Last cycle: Day 1: (T) 100mg/m2 as 1 hour IV infusion followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 22: (H) 6 mg/kg administered by IV infusion over 30 minutes.
  Interventions: Drug: docetaxel; Biological: trastuxumab
- Docetaxel, Carboplatin, and Herceptin (Experimental): Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose admin by IV over 90 mins, Day 2: Docetaxel (T) 75 mg/m2 by IV over 1 hour followed by carboplatin (C) at target AUC=6 mg/mL/min admin by IV over 30-60 mins, Day 8: (H) 2mg/kg admin by IV over 30 mins, Day 15: 2mg/kg admin by IV over 30 mins.
  Subsequent cycles: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins.
  Last cycle: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins, Day 22: (H) 6 mg/kg admin by IV over 30 mins.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: Docetaxel

INTERVENTIONS:
Biological: trastuzumab — Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose admin by IV over 90 mins, Day 2: Docetaxel (T) 75 mg/m2 by IV over 1 hour followed by carboplatin (C) at target AUC=6 mg/mL/min admin by IV over 30-60 mins, Day 8: (H) 2mg/kg admin by IV over 30 mins, Day 15: 2mg/kg admin by IV over 30 mins.
  Subsequent cycles: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins.
  Last cycle: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins, Day 22: (H) 6 mg/kg admin by IV over 30 mins.
  Other Names: herceptin
  Arms: Docetaxel, Carboplatin, and Herceptin
Drug: carboplatin — Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose admin by IV over 90 mins, Day 2: Docetaxel (T) 75 mg/m2 by IV over 1 hour followed by carboplatin (C) at target AUC=6 mg/mL/min admin by IV over 30-60 mins, Day 8: (H) 2mg/kg admin by IV over 30 mins, Day 15: 2mg/kg admin by IV over 30 mins.
  Subsequent cycles: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins.
  Last cycle: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins, Day 22: (H) 6 mg/kg admin by IV over 30 mins.
  Arms: Docetaxel, Carboplatin, and Herceptin
Drug: docetaxel — Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose administered by IV infusion over 90 minutes, Day 2: Docetaxel (T) 100 mg/m2 by IV infusion over 30 minutes, Day 8: (H) 2mg/kg administered by IV infusion over 30 minutes, Day 15: 2mg/kg administered by IV infusion over 30 minutes.
  Subsequent cycles: Day 1: (T) 100mg/m2 as 1 hour IV infusion given every 3 weeks, followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes.
  Last cycle: Day 1: (T) 100mg/m2 as 1 hour IV infusion followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 22: (H) 6 mg/kg administered by IV infusion over 30 minutes.
  Other Names: taxotere
  Arms: Herceptin plus docetaxel
Biological: trastuxumab — Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose administered by IV infusion over 90 minutes, Day 2: Docetaxel (T) 100 mg/m2 by IV infusion over 30 minutes, Day 8: (H) 2mg/kg administered by IV infusion over 30 minutes, Day 15: 2mg/kg administered by IV infusion over 30 minutes.
  Subsequent cycles: Day 1: (T) 100mg/m2 as 1 hour IV infusion given every 3 weeks, followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes.
  Last cycle: Day 1: (T) 100mg/m2 as 1 hour IV infusion followed by (H) 2 mg/kg IV infusion over 30 minutes, Day 8: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 15: (H) 2 mg/kg administered by IV infusion over 30 minutes, Day 22: (H) 6 mg/kg administered by IV infusion over 30 minutes.
  Other Names: herceptin
  Arms: Herceptin plus docetaxel
Drug: Docetaxel — Cycle 1: Day 1: Herceptin (H) 4 mg/kg loading dose admin by IV over 90 mins, Day 2: Docetaxel (T) 75 mg/m2 by IV over 1 hour followed by carboplatin (C) at target AUC=6 mg/mL/min admin by IV over 30-60 mins, Day 8: (H) 2mg/kg admin by IV over 30 mins, Day 15: 2mg/kg admin by IV over 30 mins.
  Subsequent cycles: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins.
  Last cycle: Day 1: (T) 75mg/m2 as 1 hour IV followed by (C) at target AUC=6 mg/mL/min admin by IV 30-60 mins every 3 weeks followed by (H) 2 mg/kg IV over 30 mins, Day 8: (H) 2 mg/kg admin by IV over 30 mins, Day 15: (H) 2 mg/kg admin by IV over 30 mins, Day 22: (H) 6 mg/kg admin by IV over 30 mins.
  Other Names: taxotere
  Arms: Docetaxel, Carboplatin, and Herceptin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known if docetaxel and trastuzumab are more effective with or without carboplatin in treating women who have HER2-positive breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combining docetaxel and trastuzumab with or without carboplatin in treating women who have HER2-positive stage IIIB or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to disease progression in women with HER2-positive stage IIIB, IIIC, or IV breast cancer treated with docetaxel and trastuzumab (Herceptin) with or without carboplatin.
* Compare the response rate and duration of overall response in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare rate of clinical benefit, defined as complete response, partial response, or stable disease for more than 24 weeks, in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Determine pathologic and molecular markers for predicting efficacy of these regimens in these patients.
* Determine genetic and biochemical markers for predicting risk of cardiac dysfunction and later cardiac events in patients receiving these regimens.
* Determine whether peripheral levels of shed HER2 extracellular domain constitute a prognostic and/or predictive factor of time to progression and survival of patients receiving these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to prior adjuvant and/or neoadjuvant chemotherapy (none vs with taxanes vs without taxanes) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I:

  * Course 1: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15. Patients receive docetaxel IV over 1 hour and carboplatin IV over 30-60 minutes on day 2.
  * Courses 2 and all subsequent courses: Patients receive docetaxel IV over 1 hour and carboplatin IV over 30-60 minutes on day 1 and trastuzumab IV over 30 minutes on days 1, 8, and 15.
* Arm II: Patients receive docetaxel and trastuzumab as in arm I. In both arms, treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. After completion of 8 courses, patients continue to receive trastuzumab IV over 30 minutes every 21 days in the absence of disease progression.

Patients are followed every 2 months for 3 years.

PROJECTED ACCRUAL: A total of 250 patients (125 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Stage IIIB, IIIC, or IV
  * HER2-positive
* Measurable or evaluable disease

  * Patients with osteolytic bone lesions as only site of disease must have at least 2 lytic sites confirmed by bone x-ray, MRI, or CT scan
  * None of the following are eligible as only manifestation of metastatic disease:

    * Blastic bone metastases
    * Mixed bone metastases
    * Lymphangitic carcinomatosis
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Inflammatory breast disease
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No prior or known concurrent clinical manifestation of brain or leptomeningeal involvement
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Sex

* Female

Menopausal status

* Pre- or post-menopausal

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST and ALT no greater than 5 times ULN
* Alkaline phosphatase no greater than 5 times ULN (unless due to bone metastases or any nonmalignant bone disease and in absence of liver disorders)
* AST and/or ALT greater than 1.5 times ULN AND alkaline phosphatase greater than 2.5 times ULN ineligible

Renal

* Creatinine no greater than 2 mg/dL
* Creatinine clearance at least 60 mL/min

Cardiovascular

* LVEF normal by MUGA or echocardiogram
* No myocardial infarction within the past year
* No unstable angina pectoris
* No documentation of congestive heart failure
* No concurrent grade 3 or 4 cardiovascular arrhythmia
* No poorly controlled hypertension (i.e., diastolic pressure greater than 100 mmHg)

Pulmonary

* No severe dyspnea due to complications of advanced malignancy
* No respiratory insufficiency requiring supplemental oxygen

Other

* No significant neurologic or psychiatric disorders (e.g., psychotic disorders, dementia, or seizures) that would preclude study
* No pre-existing sensory or motor neuropathy grade 2 or greater
* No other serious illness or medical condition
* No active uncontrolled infection
* No active peptic ulcer disease
* No unstable diabetes mellitus
* No other prior or concurrent malignancy except for:

  * Curatively treated nonmelanoma skin cancer
  * Carcinoma in situ of the cervix
  * Other curatively treated cancer and disease free for at least 10 years
* No known allergic reactions to study drugs
* No contraindications for the use of corticosteroids
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* No prior trastuzumab (Herceptin) for locally advanced or metastatic disease
* Prior trastuzumab-containing regimen (except with taxane) as adjuvant or neoadjuvant therapy allowed provided relapse occurred at least 6 months after therapy

Chemotherapy

* No prior chemotherapy for locally advanced or metastatic disease or local recurrence
* No prior chemotherapy with anthracycline or anthracenedione regimens with cumulative doses of more than 360 mg/m2 of doxorubicin, 720 mg/m2 of epirubicin, or 72 mg/m2 of mitoxantrone
* No prior platinum-containing regimen as adjuvant or neoadjuvant chemotherapy
* At least 4 weeks since prior anthracyclines or anthracenediones
* Prior taxanes as adjuvant or neoadjuvant chemotherapy allowed provided relapse occurred at least 6 months after therapy
* Prior taxane with trastuzumab as adjuvant or neoadjuvant chemotherapy allowed provided relapse occurred at least 12 months after therapy
* No concurrent amifostine

Endocrine therapy

* Prior hormonal therapy in the adjuvant or metastatic setting allowed provided patient has progressive disease and therapy has stopped before study entry
* Concurrent chronic corticosteroids allowed if initiated more than 6 months before study entry and at a low dose (no greater than 20 mg methylprednisolone or equivalent)
* No concurrent raloxifene, tamoxifen, or other selective estrogen receptor modulators
* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy to study lesion unless clear progression
* At least 4 weeks since prior radiotherapy (unless radiotherapy involved only a single field to treat a single metastatic bone lesion)
* Concurrent radiotherapy for palliative treatment allowed

Surgery

* Not specified

Other

* Recovered from prior antitumor therapy
* At least 30 days since prior experimental drugs
* No other concurrent experimental drugs
* No other concurrent anticancer therapy
* No concurrent bisphosphonates if osteolytic bone metastases are only site of disease

  * If receiving concurrent bisphosphonates other than for bone metastases only, must have been started at least 3 months before study entry
* No concurrent primary prophylactic antibiotics
* No concurrent cardioprotectors (e.g., dexrazoxane)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2002-05; Primary Completion 2006-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluate time to disease progression after treatment with either Herceptin in with single-agent docetaxel (TH) or Herceptin with Carboplatin and TH in metastatic breast cancer pts previously untreated with chemo whose cancer contains the HER2 gene amp. | till disease progression

SECONDARY OUTCOMES:
To compare response rate, duration of overall response, overall survival. | undefined
To evaluate and compare the rate of clinical benefit, defined as CR, PR, or stable disease > 24 weeks. | undefined
To compare toxicity between the 2 arms. | 2 years
To evaluate pathologic and molecular markers for predicting efficacy. | 2 years
Correlate peripheral levels of shed HER2 extracellular domain (ECD) with FISH results and to determine whether peripheral levels of shed HER2 ECD consitute a prognostic and/or predicitive factor vis-a-vis time to progression and survival. | undefined
To evaluate genetic and biochemical markers for predicting risk of developing cardiac dysfunction and later cardiac events in this patient population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Chap, MD, Principal Investigator — C. Klien and Associates
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Press MF, Sauter G, Bernstein L, Villalobos IE, Mirlacher M, Zhou JY, Wardeh R, Li YT, Guzman R, Ma Y, Sullivan-Halley J, Santiago A, Park JM, Riva A, Slamon DJ. Diagnostic evaluation of HER-2 as a molecular target: an assessment of accuracy and reproducibility of laboratory testing in large, prospective, randomized clinical trials. Clin Cancer Res. 2005 Sep 15;11(18):6598-607. doi: 10.1158/1078-0432.CCR-05-0636. PMID 16166438
- [Result] Pegram M, Forbes J, Pienkowski T, et al.: BCIRG 007: first overall survival analysis of randomized phase III trial of trastuzumab plus docetaxel with or without carboplatin as first line therapy in HER2 amplified metastatic breast cancer (MBC). [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA1008, 2007.
- [Result] Valero V, Roche H, Pienkowski T, et al.: BCIRG 007: serum HER2 levels in women with metastatic HER2-amplified breast cancer. [Abstract] J Clin Oncol 25 (18 Suppl 20): A-1020, 2007.
- [Result] Forbes JF, Kennedy J, Pienkowski T, et al.: BCIRG 007: randomized phase III trial of trastuzumab plus docetaxel with or without carboplatin first line in HER2 positive metastatic breast cancer (MBC): main time to progression (TTP) analysis. [Abstract] J Clin Oncol 24 (Suppl 18): A-LBA516, 7s, 2006.